CLINICAL TRIAL: NCT04355351
Title: Study of Immune Response During SARS-CoV-2 Infection
Brief Title: Study of Immune Response During SARS-CoV-2 Infection - (COVID-19)
Acronym: CovImmune
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20-PP-05
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: New Coronavirus Disease (COVID-19), Infection With SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hospital staff exposed to SARS-Cov-2 (Other)
  Interventions: Other: blood sampling
- SARS-Cov-2 infected patient (Other)
  Interventions: Other: additional blood tubes

INTERVENTIONS:
Other: blood sampling — blood sampling done on hospital staff without sars-coV-2 symptoms
  Arms: hospital staff exposed to SARS-Cov-2
Other: additional blood tubes — Additionnal blood tube taken during the classical blood sampling in hospital
  Arms: SARS-Cov-2 infected patient

SUMMARY:
Study of the cellular immune response during the SARS-CoV-2 infection and identify cytokinic profiles in caregivers exposed to the virus with asymptomatic forms of COVID19, patients with an asymptomatic form followed in ambulatory care and patients hospitalized in the infectious disease department or in resuscitation at the CHU de Nice COVID-19 according to their clinical symptomatology and the kinetics of clinical aggravation using functional tests evaluating the Th1 type immune response.

The project is divided into a clinical component comprising the study of the immune response in different populations and a cellular component focusing on the in vitro study of different immunomodulating treatments on their ability to induce an anti-viral Th1

DETAILED DESCRIPTION:
Since March 2020, Europe has been facing the spread of Coronavirus disease 2019 (COVID-19), an emerging infectious disease of viral zoonosis type, caused by the coronavirus SARS-CoV-21. This virus is responsible for an epidemic in Wuhan in November 2019 and a pandemic in March 2020. The mode of transmission, both respiratory and by contact, carried by microdroplets emitted by an infected person and inhaled by a person nearby, induces a very high contagiousness rate2. In the majority of cases, CoV-2-SARS infection is not very symptomatic, but some evolve into severe forms, particularly in frail people: elderly subjects, those affected by chronic diseases (diabetes, obesity or cancer) or those undergoing immunosuppressive treatments. There is still little information on the reasons why some will develop a severe form while others will remain asymptomatic. The immune response is little studied in this context.

Functional study of the cellular immune response has shown its interest in predicting the risk of infection in different cohorts, particularly in renal insufficiency subjects awaiting transplantation with an over-risk of developing an infection within a year in patients with a low level of gamma interferon (INFγ: main anti-viral cytokine) after non-specific stimulation of T lymphocytes.

A study published the clinical characteristics of 41 patients infected with coronavirus at the Huanan seafood market (first contact cases). Despite a similar clinical symptomatology: cough (76%) and fever (98%), some patients required rapid ventilatory assistance. These patients had an increased production of inflammatory cytokines: IL2, IL7, IL10, GSCF, IP10, MCP1, MIP1A, and TNFα3.

Here, the objective is to identify cytokine profiles in subjects exposed to or infected with SARS-CoV-2 that can predict their risk of developing a severe pauci-symptomatic form at the time of exposure or during the development of a severe form. the team believes that the immune response to this infection is a major factor in the risk of developing an asymptomatic infection, a flu-like symptomatology or a respiratory failure syndrome (ARDS).3,4 The team believes that the immune response to this infection is a major factor in the risk of developing an asymptomatic infection, a flu-like symptomatology or a respiratory failure syndrome (ARDS). The team thus wishes to better direct patients to appropriate care structures to optimise the care pathway (ambulatory, infectiology, intensive care), respirators and number of beds so as not to overload the staff) and to enable treatments to be personalised and adapted as best as possible: corticosteroids, immunomodulators, antivirals.

The study will be based on 2 axes: a first clinical axis (i) and a cellular axis (ii).

In its clinical part (i), the intensity of the immune response in COVID19 subjects presenting different forms of the disease (asymptomatic, moderate and severe forms) will be measured. These subjects will be recruited from two different patient populations:

* Subjects at risk of infection with CoV-2-SARS. We will test the Th1 response of caregivers at the time of their entry into a COVID-19 service by measuring the level of INFγ released after non-specific T-cell stimulation. The hypothesis is that a high level of INFγ at the time of exposure prevents the risk of developing severe disease and directs the patient towards less symptomatic forms. Thus, thanks to serological tests, it will be possible to determine retrospectively in this group how many subjects presented an asymptomatic form and thus to determine with the help of a functional test mimicking a viral infection the level of IFNγ measured after stimulation.
* Patients with CoV-2-SARS infection hospitalized in the Infectious Diseases Department with a moderate form or in resuscitation with a severe form of COVID.19 The evaluation of these patients on admission using a functional test mimicking a viral infection the rate of IFNγ measured after stimulation will be carried out.

The levels of IFNγ measured after stimulation will be compared in these 3 groups of COVID19 patients if the evolution towards inflammatory cytokinic profiles at D0, D5 and D10 can predict the risk of developing ARDS...

Then, the impact of different therapeutic interventions on the secretion of INFγ will be tested in vitro in an ancillary study (ii): anti-inflammatory, corticosteroids, anti-IL6, IL2, IL7, chloroquine on their capacity to produce anti-viral cytokines of the type INFγ on different T cells while limiting the production of pro-inflammatory cytokines by cells of innate immunity, from healthy subjects, COVID-19 subjects with a mildly symptomatic form or COVID-19 subjects with ARDS.

ELIGIBILITY:
1/ Medical personnel exposed to SARS-CoV-2 infection

Inclusion criteria:

* Every willing member of medical personnel who is in charge of care, treatment or transfer of patients with COVID-19, in the hospitals of Nice, Cannes and Antibes
* The absence of infection with SARS-CoV-2 at enrolment
* Age > 18 years
* Having signed an informed consent
* Valid health insurance

Non-inclusion criteria:

* Age < 18 years
* Under custody, in prison or diagnosed with a mental illness
* Refusal to give informed consent or its withdrawal
* Pregnant or breastfeeding
* Known immunodeficiency
* Previous immunosuppressive therapy

  2) Subjects hospitalized for a SARS-CoV-2 infection

Inclusion criteria:

* All adult patients hospitalized in the intensive care or in infectious diseases units, or receiving follow-up at the dermatology unit, in Nice University Hospital, diagnosed with COVID-19 (as defined by the positivity to SARS-CoV-2 by two PCR multiplex)
* Age > 18 years
* Having signed an informed consent

Non-inclusion criteria:

* Age < 18 years
* Under custody, in prison or diagnosed with a mental illness
* Refusal to give informed consent or its withdrawal
* Pregnant or breastfeeding
* Known immunodeficiency
* Previous immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2021-12-04 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Level of IFN-gamma after a non-specific stimulation of T lymphocytes | 6 months
  Peripheral T lymphocytes will be stimulated with an anti-CD3 for 16-24h. The Level of IFN-gamma (pg/mL) will be defined using an automated ELISA test (Protein Simple) on the stimulated and non-stimulated plasma.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Antibes Hospital, Antibes
  - Cannes Hospital, Cannes
  - Nice Hospital, Nice

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buscot M, Cremoni M, Graca D, Brglez V, Courjon J, Allouche J, Teisseyre M, Boyer L, Barriere J, Chamorey E, Carles M, Seitz-Polski B. Breakthrough infections due to SARS-CoV-2 Delta variant: relation to humoral and cellular vaccine responses. Front Immunol. 2023 Mar 30;14:1145652. doi: 10.3389/fimmu.2023.1145652. eCollection 2023. PMID 37063916